CLINICAL TRIAL: NCT01868880
Title: Effect of Heart Rate Control Using Ivabradine and Beta-blockers Combination Versus Beta-blockers Up-titration on Ventricular Pacing in Heart Failure Patients With an Implanted Cardioverter Defibrillator.
Brief Title: Effect of Ivabradine and Beta-blockers Combination Versus Beta-blockers Up-titration on Right Ventricular Pacing
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulties in recruiting patients
Sponsor: Policlinico Casilino ASL RMB (Other)
Responsible Party: Principal Investigator, Leonardo Calò, MD, MD, FESC, Policlinico Casilino ASL RMB
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: calo03; calo03 (Other: Policlinico Casilino)
Record Dates: First submitted 2013-05-09; First posted 2013-06-05 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Heart Rate Control in ICD Patients With Heart Failure
MeSH Terms: interventions — Ivabradine; Adrenergic beta-Antagonists; Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ivabradine plus beta-blocker(bisoprolol) (Experimental): Ivabradine will be administered at a dose of 5 mg twice daily in addition to a low dose of beta-blocker (bisoprolol 1,25 or 2,5 mg). After four weeks of treatment ivabradine will be eventually lowered up to 2,5 mg twice daily in the presence of side effects (phosphenes, diplopia, headache or dizziness).
  Interventions: Drug: Ivabradine plus beta-blocker (bisoprolol)
- beta-blocker (bisoprolol) titration (Active Comparator): Beta blocker Bisoprolol will be titrated biweekly starting from the initial dose of 1,25-2,5 mg daily up to the max dose of 10 mg daily or to the maximum tolerated dose.
  Interventions: Drug: betablocker titration

INTERVENTIONS:
Drug: Ivabradine plus beta-blocker (bisoprolol) — Ivabradine will be administered at a dose of 5 mg twice daily in addition to a low dose of beta-blocker (bisoprolol 1,25 or 2,5 mg). After four weeks of treatment ivabradine will be eventually lowered up to 2,5 mg twice daily in the presence of side effects (phosphenes, diplopia, headache or dizziness).
  Arms: ivabradine plus beta-blocker(bisoprolol)
Drug: betablocker titration — Beta blocker Bisoprolol will be up-titrated biweekly starting from the initial dose of 1,25-2,5 mg daily up to the max dose of 10 mg daily or to the maximum tolerated dose.
  Arms: beta-blocker (bisoprolol) titration

SUMMARY:
The aim of this prospective, randomized and controlled trial is to evaluate the use of the ivabradine in combination to a low-dose of beta-blocker (bisoprolol) versus up-titration of beta-blocker (bisoprolol) to obtain heart rate (HR) control with reduction in RV pacing in single-chamber or dual chambers ICD recipients HF patients with moderate to severe left ventricular dysfunction (FE ≤ 40%) and an heart rate ≥ 70 bpm in sinus rhythm over a 12-months follow up.

Besides the investigators want to assess if the combination of ivabradine to a low-dose of beta-blocker (bisoprolol) versus up-titration of beta-blocker (bisoprolol) may determine a lower degree of left ventricular dysfunction progression, the reduction of ventricular arrhythmias burden and ICD appropriate therapy occurrence and the improvement of quality of life in ICD heart failure patients.

DETAILED DESCRIPTION:
Background

High heart rate (HR) represent per se a risk factor for cardiovascular mortality and heart failure (HF) progression, despite optimal HF therapy. Beta-blockers remain the therapy of choice in all patients with systolic HF, but they may worsen atrioventricular (AV) conduction and increase right ventricular (RV) pacing percentage. Several studies have demonstrated detrimental effects of RV pacing on cardiac function. Percent RV pacing > 40-50% is an independent predictor of death and hospitalization for HF in implantable cardioverter-defibrillator(ICD) patients, particularly in those with preexistent left ventricular dysfunction.1,2 Cumulative RV pacing > 2% and ejection fraction (EF) < 40% are independent predictors for Ventricular Tachycardia(VT)/Ventricular Fibrillation (VF) occurrence in ICD patients.3 Therefore reduction of cumulative RV pacing as far as possible should be achieved in ICD patients. Ivabradine is a specific inhibitor of the If current of the sinus node, that induces a selective and dose dependent HR reduction; it is a pure HR lowering agent without effects on AV conduction or contractility.4 In HF patients implanted with an ICD ivabradine could act as an heart rate control drug in combination with a beta-blocker without increase right ventricular (RV) pacing percentage and may be an option to reduce left-ventricular dysfunction progression and ventricular arrhythmias burden and appropriate ICD therapy.

Aim

The aim of this prospective, randomized and controlled trial is to evaluate the use of the ivabradine in combination to a low-dose of beta-blocker (bisoprolol) versus up-titration of beta-blocker (bisoprolol) to obtain heart rate (HR) control with reduction in RV pacing in single-chamber or dual chambers ICD recipients HF patients with moderate to severe left ventricular dysfunction (FE ≤ 40%) and an heart rate ≥70 bpm in sinus rhythm over a 12-months follow up.

Besides we want to assess if the combination of ivabradine to a low-dose of beta-blocker (bisoprolol) versus titration of beta-blocker (bisoprolol) may determine a lower degree of left ventricular dysfunction progression, the reduction of ventricular arrhythmias burden and ICD appropriate therapy occurrence and the improvement of quality of life in ICD heart failure patients.

Endpoints of the study

Primary endpoints:

Right ventricular pacing percentage increase > 50% or Cardiovascular death or Heart failure decompensation or Crossover due to worsening heart failure.

Secondary endpoints:

Ejection fraction decrease < 5% and Left Ventricular End-Systolic Volume decrease <15%.

Ventricular arrhythmias and ICD appropriate therapy reduction. Heart rate variability improvement NYHA Classification improvement Minnesota Living With Heart Failure Questionnaire (MLHFQ) total score reduction.

Right ventricular pacing percentage. Composite endpoint: cardiovascular death and hospitalization due to worsening heart failure.

Crossover rate due to worsening heart failure

Study protocol:

Baseline assessment:

Clinical visit: demographic data, risk factors for cardiovascular disease, primary cause of heart failure, NYHA class, comorbidities, echocardiographic parameters, drug therapy, cardiovascular hospitalizations in the last year.

Rest ECG (for assessment of rest heart rate, presence of sinus rhythm or device-induced rhythm, QRS duration); Blood pressure measurement; Electronic device control (for assessment of right ventricular stimulation percentage; electrical parameters and arrhythmias diagnostic data); Echocardiogram (for assessment of left ventricular end-diastolic and end-systolic volumes, left ventricular ejection fraction); MLHFQ

Assignment of consecutive patients to treatment with ivabradine plus beta-blocker(bisoprolol) or beta-blocker (bisoprolol) titration. Mean Heart Rate Target is 55-70 bpm for both groups.

Ivabradine will be administered at a dose of 5 mg twice daily in addition to a low dose of beta-blocker (bisoprolol 1,25 or 2,5 mg). After four weeks of treatment ivabradine will be eventually lowered up to 2,5 mg twice daily in the presence of side effects (phosphenes, diplopia, headache or dizziness).

Beta blocker Bisoprolol will be up-titrated biweekly starting from the initial dose of 1,25-2,5 mg daily up to the max dose of 10 mg daily or to the maximum tolerated dose.

Patients are controlled in office follow-up visits after 3, 6 and 12 months, in addition to a Remote Monitoring program for clinical data and trend reviewing at least every 15 days or as soon as possible whenever a Remote Monitoring alert notification is received. Besides every 15 days patients will receive a telephone contact in order to evaluate their clinical state and to uptitrate the beta blocker therapy based on mean heart rate detected trough remote control of the ICD.

Three months in-office follow-up:

Clinical visit: symptoms, NYHA class, drug therapy, cardiovascular hospitalizations in the last three months.

Rest ECG (for assessment of rest heart rate, presence of sinus rhythm or device-induced rhythm, QRS duration); Blood pressure measurement; Echocardiogram (for assessment of left ventricular end-diastolic and end-systolic volumes, left ventricular ejection fraction); Electronic device control (for assessment of right ventricular stimulation percentage; electrical parameters and arrhythmias diagnostic data) .

Six months in office follow-up:

Clinical visit: NYHA class, comorbidities, echocardiographic parameters, drug therapy, cardiovascular hospitalizations in the last three months.

Rest ECG (for assessment of rest heart rate, presence of sinus rhythm or device-induced rhythm, QRS duration); Echocardiogram (for assessment of left ventricular end-diastolic and end-systolic volumes, left ventricular ejection fraction); Electronic device control (for assessment of right ventricular stimulation percentage; electrical parameters and arrhythmias diagnostic data).

MLHFQ

One year in office follow-up:

Clinical visit: NYHA class, comorbidities, echocardiographic parameters, drug therapy, cardiovascular hospitalizations in the last three months.

Rest ECG (for assessment of rest heart rate, presence of sinus rhythm or device-induced rhythm, QRS duration); Electronic device control (for assessment of right ventricular stimulation percentage; electrical parameters and arrhythmias diagnostic data).

Echocardiogram (for assessment of left ventricular end-diastolic and end-systolic volumes, left ventricular ejection fraction); MLHFQ

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years.

Patients with stable chronic heart failure implanted with mono-cameral or bicameral ICD with a home monitoring remote control.

Moderate to severe left ventricular dysfunction (FE ≤ 40%).

Any cause of heart failure was allowed apart congenital heart disease.

Bicameral ICD programmed in DDD or AAI/DDD with AV interval < 300 msec.

Rest ECG heart rate ≥70 bpm;

Sinus rhythm.

In therapy with low-dose of beta-blocker (bisoprolol 1,25-2,5 mg) and with the maximum dose tolerated of angiotensin-converting enzyme inhibitor or blockade of angiotensin II receptor, mineralocorticoid antagonist, antiplatelet and lipid-lowering therapy, unless contraindicated.

Exclusion Criteria:

Inability of providing informed consent;

Age < 18 years.

State of pregnancy or lactation.

Recent (<2 months) myocardial infarction;

Contraindications to beta-blockers and ivabradine;

Rest ECG heart rate < 70 bpm;

No sinus rhythm.

Administration of non-dihydropyridinic calcium channels antagonists, digitalis, class I antiarrhythmic drugs, strong inhibitors of cytochrome P450 3A4 at the time of enrollment.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Right ventricular pacing percentage increase > 50% or cardiovascular death or Heart failure decompensation or Crossover due to worsening heart failure. | 12 months

SECONDARY OUTCOMES:
Number of episodes of non-sustained and sustained ventricular tachycardia and ventricular fibrillation | 12 months
Number of ICD shock-delivery for ventricular fibrillation and sustained ventricular tachycardia | 12 months
Ejection fraction decrease < 5% from baseline value | 12 months
Left Ventricular End-Systolic Volume decrease <15% from baseline value | 12 months
Heart rate variability increase (> 10%) from baseline value | 12 months
reduction of at least one NYHA Class from baseline value | 12 months
Change in Minnesota Living Heart Failure Questionnaire scores (>5) from the baseline score. | 12 months
Right ventricular pacing percentage reduction (> 10%) from baseline value | 12 months
Composite endpoint: number of cardiovascular death and hospitalization due to worsening heart failure. | 12 months
Crossover rate due to worsening heart failure | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Polinico Casilino, Rome, Italy

REFERENCES:
- [Background] Sharma AD, Rizo-Patron C, Hallstrom AP, O'Neill GP, Rothbart S, Martins JB, Roelke M, Steinberg JS, Greene HL; DAVID Investigators. Percent right ventricular pacing predicts outcomes in the DAVID trial. Heart Rhythm. 2005 Aug;2(8):830-4. doi: 10.1016/j.hrthm.2005.05.015. PMID 16051118
- [Background] Smit MD, Van Dessel PF, Nieuwland W, Wiesfeld AC, Tan ES, Anthonio RL, Van Erven L, Van Veldhuisen DJ, Van Gelder IC. Right ventricular pacing and the risk of heart failure in implantable cardioverter-defibrillator patients. Heart Rhythm. 2006 Dec;3(12):1397-403. doi: 10.1016/j.hrthm.2006.08.006. Epub 2006 Aug 10. PMID 17161779
- [Background] Borer JS, Le Heuzey JY. Characterization of the heart rate-lowering action of ivabradine, a selective I(f) current inhibitor. Am J Ther. 2008 Sep-Oct;15(5):461-73. doi: 10.1097/MJT.0b013e3181758855. PMID 18806523